CLINICAL TRIAL: NCT07096622
Title: Efficacy of Visual and Perceptual Training on Visual Function for Operative Congenital Ectopia Lentis Children: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Visual and Perceptual Training on Visual Function for Operative Congenital Ectopia Lentis Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Guangming Jin, Associate Chief Physician, Cataract Department, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025KYPJ068
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Ectopia Lentis; Lens Subluxation or Dislocation
MeSH Terms: conditions — Ectopia Lentis; Lens Subluxation

STUDY DESIGN:
Intervention Model Description: Open-label, single-center, parallel-group randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This study employs an open-label design without participant or investigator blinding, but with assessor blinding implemented. To reduce bias under non-blinded conditions, trial-related personnel involved in participant screening remain blinded, and clinical staff conducting regular ophthalmological examinations and data analysts are kept blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in the intervention group should undergo a re-examination at baseline and be fitted with appropriately prescribed glasses based on the examination results, which should be worn throughout the day; After receiving guidance from a trainer, participants will undergo treatment using the visual perception training therapy software (HVT, version number: V1.0.10000) on the online platform, for 30 minutes daily, over a total period of 3 months. Follow-up visits and eye examinations will be conducted at the 1st, 2nd, and 3rd months following the start of the trial.
  Interventions: Device: perceptual learning visual treatment,HVT
- compare group (No Intervention): Participants in the control group should undergo a re-examination at baseline, select glasses with appropriate prescriptions based on the examination results, wear them throughout the day, and continue for a total of 3 months. Follow-up visits and eye examinations will be conducted at 1, 2, and 3 months after the start of the trial.

INTERVENTIONS:
Device: perceptual learning visual treatment,HVT — After receiving guidance from a trainer, treatment was conducted using the visual perception training therapy software (HVT, version number: V1.0.10000) on a network platform for 30 minutes per day, totaling 3 months.
  Arms: intervention group

SUMMARY:
This is a single-centre, open-label, parallel-group randomized controlled trial with the following objectives: Firstly, the investigators aim to evaluate the efficacy of web-based visual and perceptual training therapy on visual function in children with postoperative congenital ectopia lentis. Secondly, the investigators target to investigate the proportion of patients achieving ≥2 lines improvement in best-corrected visual acuity (BCVA), changes in stereoacuity, quality of life scores, and treatment compliance following visual and perceptual training intervention. Thirdly, to explore the safety profile of visual and perceptual training therapy software in this specific patient population. Lastly, this study aims to provide evidence-based recommendations for visual rehabilitation training strategies in children with postoperative congenital ectopia lentis in the Chinese population.

DETAILED DESCRIPTION:
Congenital ectopia lentis (CEL) is commonly observed in patients with Marfan syndrome. It is a rare genetic eye disorder caused by abnormal development of the lens zonules, leading to displacement of the lens from its normal anatomical position. In addition to abnormalities in the development of refractive media such as the cornea and lens, these patients may also exhibit abnormalities in the photoreceptive system, including the retina. Furthermore, since the patients receive abnormal visual input stimuli during the critical period of visual development, this often leads to the development of amblyopia in both eyes. Currently, for patients with severe visual impairment due to lens dislocation, the standard treatment involves lens extraction combined with primary intraocular lens implantation. However, for patients with bilateral amblyopia following CEL surgery, conventional treatment involves full-time refractive correction, which cannot prevent residual amblyopia. Additionally, patients who undergo extracapsular artificial lens implantation may experience astigmatism due to potential lens tilt post-surgery, which can impair visual function and mental health.

Visual perception training therapy (HVT) is an emerging treatment modality for amblyopia. Studies have shown that compared to traditional refractive correction and occlusion therapy, visual perception training therapy offers faster visual acuity improvement, higher compliance, and the ability to enhance binocular visual function. Furthermore, existing research indicates that for patients with anisometropia or small-angle strabismic amblyopia, the efficacy of visual perception training therapy combined with refractive correction is superior to refractive correction alone. As a form of visual perception training therapy software, web-based visual perception training therapy enables patients to complete training at home through game-based activities. It can also adjust training plans based on patients' conditions and training progress, offering personalized treatment plans to enhance treatment compliance and patient experience while enabling remote management by hospitals. The meridian perception learning module is particularly effective in improving uncorrected visual function for patients with astigmatism undergoing CEL surgery. However, to date, no studies have focused on the efficacy of visual perception training therapy in improving visual function for this specific population of CEL postoperative patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4-12 years, regardless of gender;
2. Previously diagnosed with congenital ectopia lentis;
3. History of bilateral lens extraction combined with intraocular lens suspension surgery, with the second eye surgery completed within 1 month ± 1 week;
4. Bilateral best-corrected visual acuity no less than 20/200 but below age-appropriate normal levels: for 4-year-old children, bilateral best-corrected visual acuity no better than 20/40; for children aged 5 years and above, bilateral best-corrected visual acuity no better than 20/30;
5. Written informed consent signed by both patients and parents/guardians.

Exclusion Criteria:

**Exclusion Criteria:**

1. History of ocular trauma or previous ocular surgery;
2. Unable to cooperate with treatment, examination, or follow-up assessments;
3. Concurrent lens dislocation recurrence, severe cataracts (dense, located on the visual axis, opacity diameter >3mm affecting central vision), secondary glaucoma, corneal endothelial decompensation, or retinal detachment requiring urgent surgical intervention;
4. Presence of diplopia in either eye;
5. Known history of neurological disorders (such as photosensitive epilepsy);
6. Post-operative participation in other clinical trials that may affect the results of this study;
7. Use of local/systemic medications that may cause visual impairment or other visual treatments (such as atropine eye drop suppression therapy, occlusion therapy, digital therapy, Bangerter filters, optical suppression, VR training, etc.) other than refractive correction within the past 3 months.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in BCVA relative to baseline in both eyes | From start of intervention to the end of intervention at 3 months
  The best corrected vision will be measured by a professional optometrist.

SECONDARY OUTCOMES:
Proportion of eyes with a relative improvement in BCVA of ≥2 lines from baseline | From start of intervention to the end of intervention at 3 months
  The best corrected vision will be measured by a professional optometrist.
Changes in stereoscopic vision relative to the baseline | From start of intervention to the end of intervention at 3 months
  Measure near stereopsis using the BUTTERFLY STEROTEST's STEREOTEST-ANIMALS part at 40 cm（16 inches） distance, wearing a pair of Standard 3-D Viewers.The angle of stereopsis of participants will be classified to 400 seconds,200 seconds and 100 seconds if they could recognize the 3-D cat, rabbit or monkey.
Change in quality of life score | From start of intervention to the end of intervention at 3 months
  This study used the PedsQL 4.0 Chinese version questionnaire to assess participants' quality of life at baseline, fisrt month, second month and third month. Participants will be asked to finish this questionnaire in paper.
  Participants aged 4 years should have their parents complete the questionnaire on their behalf. Participants aged 5-7 years should have the questionnaire completed by the researcher based on the child's responses after questioning the child. Participants aged 8-12 years should complete the questionnaire themselves. When participants did not understand the meaning of the questionnaire or had questions about the options, the researcher or parent should explain it to them and assist them in completing the questionnaire.
adherence of intervention | From start of intervention to the end of intervention at 3 months
  Compliance with refractive correction is recorded in the case report form through self-reporting at each follow-up visit.
  Compliance with visual perception training therapy software (HVT) will be automatically monitored through the system backend.
  Compliance with refractive correction will be calculated by dividing the average actual time spent wearing glasses per day over the past week, as recalled by participants during follow-up, by the average time spent awake per day, multiplied by 100%. Compliance with visual perception training will be calculated by dividing the actual number of days participants completed the training during follow-up by the number of days since the intervention began, multiplied by 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Guangming Jin, M.D., Principal Investigator — Guangdong Provincial Clinical Research Center for Ocular Diseases, State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangdong Provincial Key Laboratory of Ophthalmology and Visual Science, Guangzhou, Guangdong; Zhenzhen Liu, M.D., Study Chair — Guangdong Provincial Clinical Research Center for Ocular Diseases, State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangdong Provincial Key Laboratory of Ophthalmology and Visual Science, Guangzhou, Guangdong; Danying Zheng, M.D., Study Chair — Guangdong Provincial Clinical Research Center for Ocular Diseases, State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangdong Provincial Key Laboratory of Ophthalmology and Visual Science, Guangzhou, Guangdong
Locations (1):
- Guangdong Provincial Clinical Research Center for Ocular Diseases, State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangdong Provincial Key Laboratory of Ophthalmology and Visual Science, Guangzhou, Guangdong, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and results will be published in a peer-reviewed journal.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available on December 2030 for 10 years.
Access Criteria: Data are available upon reasonable request by contacting with the corresponding author.

REFERENCES:
- [Background] Yao Y, He Y, Wen Y, Feng L, Ye Q, Xu Z, Zhou Y, Pang Y, Yu W, Zhong Y, Li Q, Yuan J, Liu J, Li J. Factual Evidence on Digital Therapeutics in Pediatric Amblyopia: Insights into Rapid Axial Elongation Risk. Ophthalmology. 2025 Jun;132(6):661-670. doi: 10.1016/j.ophtha.2025.01.005. Epub 2025 Jan 13. PMID 39814322
- [Background] Xiao S, Angjeli E, Wu HC, Gaier ED, Gomez S, Travers DA, Binenbaum G, Langer R, Hunter DG, Repka MX; Luminopia Pivotal Trial Group. Randomized Controlled Trial of a Dichoptic Digital Therapeutic for Amblyopia. Ophthalmology. 2022 Jan;129(1):77-85. doi: 10.1016/j.ophtha.2021.09.001. Epub 2021 Sep 14. PMID 34534556
- [Background] Liu Z, Lin H, Jin G, Tan X, Qu B, Jin L, Chen X, Wang W, Han X, Xu J, Ying G, Han Y, He M, Congdon N, Chen W, Luo L, Liu Y. In-the-Bag Versus Ciliary Sulcus Secondary Intraocular Lens Implantation for Pediatric Aphakia: A Prospective Comparative Study. Am J Ophthalmol. 2022 Apr;236:183-192. doi: 10.1016/j.ajo.2021.10.006. Epub 2021 Oct 13. PMID 34653355
- [Background] Chen T, Deng M, Zhang M, Chen J, Chen Z, Jiang Y. Visual outcomes of lens subluxation surgery with Cionni modified capsular tension rings in Marfan syndrome. Sci Rep. 2021 Feb 4;11(1):2994. doi: 10.1038/s41598-021-82586-6. PMID 33542371
- [Background] Jia WN, Chen ZX, Wang YL, Shen X, Chen XY, Chen TH, Sun Y, Liu Y, Song LH, Huo QY, Jiang YX. Genotype Associated With Visual Prognosis in Patients With Congenital Ectopia Lentis Following Lens Surgery: A Prospective Cohort Study. Am J Ophthalmol. 2024 Dec;268:285-295. doi: 10.1016/j.ajo.2024.08.002. Epub 2024 Aug 8. PMID 39121940
- [Background] Ng K, Xu P, Jin G, Cheng W, Luo X, Ding X, Zheng D, Liu Y. Quantitative analysis of choriocapillaris flow deficits and choroidal thickness in children with Marfan syndrome. Br J Ophthalmol. 2024 Jan 29;108(2):274-279. doi: 10.1136/bjo-2022-322535. PMID 36575623
- [Background] Huo QY, Zhang RZ, Jia WN, Wang YL, Shen X, Chen XY, Chen TH, Liu Y, Song LH, Wang X, Lv Y, Chen ZX, Jiang YX. Corneal Biomechanics Are Associated With FBN1 Mutations in Patients With Marfan Syndrome and Ectopia Lentis. Invest Ophthalmol Vis Sci. 2025 Mar 3;66(3):23. doi: 10.1167/iovs.66.3.23. PMID 40062814